CLINICAL TRIAL: NCT02051920
Title: Measurement of Cardiac Elastography: an Intraoperative Cardiac Surgery Study. Cardiac Elastography in Vivo
Brief Title: Cardiac Elastography Measurement : an Intraoperative Cardiac Surgery Study
Acronym: REA-FO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: REA-FO-2013-A00593-42
Record Dates: First submitted 2013-10-25; First posted 2014-01-31 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Diastolic Dysfunction and Cardiac Stiffness
Keywords: Elastography

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Since 20 years, the techniques of direct measurement of cardiac stiffness in the diagnosis of myocardial diseases do not exist.

We propose a human study evaluating the direct measurement of cardiac ultrasound stiffness by elastography.

This study will include 30 patients with cardiac disease whose rigidity varies with underlying disease.

The purpose of this study is to evaluate the stiffness during open heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Patients older than 18 years
* Every patient scheduled for cardiac surgery
* Cardiac catheterization within 6 months before surgery,
* Women of childbearing age in effective contraception (a urine pregnancy test will be performed)
* Patient affiliated or covered by a plan of health insurance.
* Francophone

Exclusion Criteria:

* Pregnant or lactating woman,
* Functional walking disability,
* Patient placed under judicial protection: guardianship,
* Patient participating in another trial and / or participated in another trial within two months,
* Patient under guardianship or trusteeship,
* Women who are not effective contraception,
* Patient with no liberty by administrative or judicial decision

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Young's Modulus measurement according to the equation E = Young 3ρCs ² | During herat surgery (Day 0)
  Ultrasound acquisition will be completed in epicardial vue using a linear probe SuperLinear 15-4 ™ connected to an ultrasound (AixplorerTM ® from Supersonic Imagine). The acquisitions will be completed in mode B + Elastrography Shear Wave ™ (SWE). A sterile gel is deposited in the bottom of the pouch of sterile protection of the probe. Many measurements will be done on accessible left and right ventricle areas.
  Measurement of Young's modulus: automated by the onboard model according to the equation E = Young 3ρCs ², where E is the Young's elastic modulus software, ρ is the tissue density and Cs the velocity of shear wave

SECONDARY OUTCOMES:
diastolic function parameters | Day 0
  Correlation between young's modulus and diastolic function parameters is assess after surgery by post processing

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Bauer, MD,PhD, Study Director — University Hospital, Rouen
Locations (1):
- Caen University Hospital, Caen, Basse Normandie, France